CLINICAL TRIAL: NCT02349568
Title: The Cost Effectiveness Between EUS-based Strategy Versus Endoscopic Retrograde Cholangiopancreatography ( ERCP )-Based Strategy in Diagnosis of Common Bile Duct Stones in Patients With Intermediate Risk: a Study in Developing Country.
Brief Title: The Cost Effectiveness of Endoscopic Ultrasound ( EUS ) Based Strategy in Diagnosis of Common Bile Duct Stones
Status: Completed | Type: Observational
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Nisa Netinatsunton, NKC Institute of Gastroenterology and Hepatology, Prince of Songkla University
Other Study IDs: EC-55-066-21-1-2
Record Dates: First submitted 2015-01-16; First posted 2015-01-29 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: Common Bile Duct Calculi
MeSH Terms: conditions — Gallstones

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- High risk group: High risk group was defined when CBD stones was detected by ultrasound ( US ) / computed tomography ( CT ) or dilated duct with abnormal LFT.
  Interventions: Procedure: High risk group
- Intermediate risk group: Intermediate risk group was defined when US/CT showed normal bile duct with abnormal LFT or dilated duct with normal LFT.
  Interventions: Procedure: Intermediate risk group

INTERVENTIONS:
Procedure: High risk group — Patients with high risk underwent EUS examination under conscious sedation. EUS was examined from second part of duodenum up to duodenal bulb. All patients even if negative EUS examination of CBD stone were underwent ERCP in the same session. The ERCPs were performed in standard manner. All patients were contacted by phone on day 1, 3 and 30 after the procedure.
  Other Names: EUS examination follow by ERCP
  Groups: High risk group
Procedure: Intermediate risk group — Patients with intermediate risk underwent EUS examination under conscious sedation. EUS was examined from second part of duodenum up to duodenal bulb. ERCPs were done at the discretion of the attending physicians. The ERCPs were performed in standard manner. The patients without ERCP done were contacted at 3 months interval to assess symptoms and LFT for 12 months.
  Other Names: EUS examination follow by ERCP or clinical follow up
  Groups: Intermediate risk group

SUMMARY:
Multiple reports in the literature showed the efficacy of EUS comparable to ERCP in the diagnosis of common bile duct ( CBD ) stone. The EUS-based strategy has provided the cost effectiveness in diagnosis of CBD stone in defined patient risk groups was showed in previous studies. The aim of our study was to assess the cost effectiveness of EUS based strategy versus ERCP based strategy in diagnosis of CBD stones in patients with intermediate risks for CBD stones in a real working situation in a developing country.

DETAILED DESCRIPTION:
Background: Multiple reports showed the efficacy of EUS comparable to ERCP in the diagnosis of CBD stone. The EUS-based strategy has provided the cost saving in diagnosis of CBD stone in patients with intermediate risk in previous studies in western population. There were multiple parameters involved the cost effectiveness analysis included cost of ERCP, cost of EUS, prevalence of CBD stones, the sensitivity and specificity of EUS and the rate of complications related to EUS and ERCP. These parameter may vary from center to center and from region to region.

Aims: To assess the cost effectiveness of EUS based strategy versus ERCP based strategy in diagnosis of CBD stones in patients with intermediate risk in a developing country.

Method : A prospective study in 141 patients with suspected CBD stones based on clinical, biochemical and imaging by trans-abdominal ultrasonography or computed abdominal tomography. All patients underwent EUS. All patients with high risk for CBD stone underwent ERCP after the EUS. For patients with intermediate risk for CBD stone, ERCP's were done at the discretion of the attending physicians. For patients with ERCP done, the diagnosis of CBD stone was confirmed by ERCP demonstration of CBD stone. In patients with intermediate risk without ERCP done, clinical follow up to assess biliary symptoms and liver function test as surrogated markers for CBD stone at 3 months interval for one year were done. The false negative rate in patients with EUS and ERCP done in this study was used to estimate the false negative rate in patients in clinical surrogated group.

Definition: High risk of CBD stones was defined when CBD stone was detected by US/CT or dilated duct with abnormal liver function test ( LFT ). Intermediate risk of CBD stones was defined when US/CT showed normal bile duct with abnormal LFT or dilated duct with normal LFT.

Cost analysis :The cost of making diagnosis of CBD stone excluding all costs of treatment was analyzed. The cost of all patients with suspected CBD stones undergoing ERCP was calculated and compared with the strategy of EUS follow by ERCP. The cost was evaluated by (1) mean costs of EUS and ERCP based on the actual cost in our center which included costs of medical staffs, disposable materials, drugs, equipment amortization and maintenance. (2) cost associated with complications induced by the procedure.

Statistical analysis: Test performance of the endoscopic ultrasound in diagnosis of CBD stones was analyzed with two by two tables. The sensitivity, specificity, positive and negative predictive values were calculated.

ELIGIBILITY:
Inclusion Criteria:

* history of biliary pain or recent cholangitis
* acute pancreatitis
* abnormal liver function test
* dilatation of CBD and or CBD stone detected by trans-abdominal ultrasound and or computed tomography.

Exclusion Criteria:

* unstable hemodynamics
* severe coagulopathy
* refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with suspected CBD stones based on clinical, biochemical and imaging by trans-abdominal ultrasonography or computed tomography..
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2012-05; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The cost of making diagnosis of CBD stone | within 12 months after EUS
  The cost of making diagnosis of CBD stone will be measured as the difference in the cost of all patients undergoing ERCP and ERCP follow by EUS intervention. The cost was evaluated by (1) mean costs of EUS and ERCP based on the actual cost in our center which included costs of medical staffs, disposable materials, drugs, equipment amortization and maintenance. (2) costs associated with complications induced by the procedure.

SECONDARY OUTCOMES:
The accuracy of EUS in diagnosis of CBD stone | within 12 months after EUS
  This will be measured as proportion of patients who encounter a correctly diagnosis of CBD stone by EUS. Positive EUS finding was confirmed by ERCP. Negative EUS finding was confirmed by ERCP or absence of symptoms for 12 months.
The safety of EUS and ERCP procedure | within 1 months
  This will be measured as proportion of patients who encounter a procedural complication (%) during EUS and ERCP that includes pancreatitis, perforation or hemorrhage

CONTACTS AND LOCATIONS:
Overall Officials: Bancha Ovartlarnporn, MD, Study Director — NKC Institue of Gastroenterology and Hepatology, Faculty of Medicine, Prince of Songkla University, Hatyai, Songkla, Thailand.
Locations (1):
- NKC Institues of Gastroenterology and Hepatology, Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand